CLINICAL TRIAL: NCT05179707
Title: A Prospective, Multicenter Research for Combination of Prostate Health Index (Phi) and mpMRI PI-RADS in the Diagnosis of Prostate Cancer
Brief Title: A Research for Combination of Prostate Health Index (Phi) and mpMRI PI-RADS in the Diagnosis of Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Zibo Central Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: CSZ01
Record Dates: First submitted 2021-12-01; First posted 2022-01-05 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Before prostate puncture, the patient's serum was collected for PHI detection, and multi-parameter MRI was performed to obtain the PI-RADS score. The sensitivity and specificity of PHI combined with PI-RADS score in the diagnosis of clinically significant prostate cancer were explored.

DETAILED DESCRIPTION:
This study is a multi-center prospective study. Patients who meet the indications for prostate puncture and whose PSA is in the gray area (4.0~10.0 ng/mL) undergo standard prostate biopsy. The patient's serum was collected for PHI detection before puncture, and multi-parameter MRI was performed before puncture. To explore the sensitivity and specificity of PHI combined with PI-RADS score in the diagnosis of clinically meaningful prostate cancer. Assess the benefit of combining PHI and mpMRI before biopsy compared with phi or mpMRI alone. Formulate clinical recommendations for PHI and mpMRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected prostate cancer
* Patients can perform standardized prostate biopsy

Exclusion Criteria:

* Have a history of prostate cancer
* Use of drugs that affect PSA before blood sampling

Ages: 50 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Male patients aged 50 to 80 years with indications for prostate puncture
Sampling Method: Probability Sample
Enrollment: 936 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Prostate Health Index | 1 year
  PHI is a simple, FDA-approved blood test that helps determine the probability of detecting prostate cancer with a biopsy. This test uses an algorithm to assess total PSA, free PSA, and p2PSA,
PI-RADS score | 1 year
  In PI-RADS, based on the comprehensive manifestations of prostate T2WI, DWI and DCE, a scoring method is given for the possibility of clinically significant prostate cancer. Specifically: 1 point: very low, extremely unlikely to exist; 2 points: low, impossible to exist; 3 points: moderate, suspicious existence; 4 points: high, may exist; 5 points: very high, extremely likely to exist.
Prostate biospy pathology | 1 year
  The pathological results of prostate puncture are used as the gold standard for the diagnosis of prostate cancer, indicating whether the patient is really suffering from prostate cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shandong, China